CLINICAL TRIAL: NCT06596707
Title: Comparison of Proximal Contact Tightness of Zirconia Reinforced Glass Ionomer Versus Conventional Nanohybrid Resin Composite: a Randomized Clinical Trial
Brief Title: Contact Tightness of Zirconomer Versus Nanohybrid Composite in Occlusoproximal Cavities in Molars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Fathi Abdelsalam, Principal in investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2255884
Record Dates: First submitted 2023-08-25; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Contact Tightness in Restoring Proximal Surfaces in Posterior Teeth
Keywords: Zirconomer; Glass Ionomer; Contact tightness; Occlusoproximal cavities; Resin composite; Class II

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zirconomer in Class II cavities (Experimental): Zirconia modified glass ionomer restorative material
  Interventions: Procedure: Zirconomer
- Nanohybrid composite in Class II cavities (Active Comparator): Conventionally used aesthetic restorations in class II
  Interventions: Procedure: Nanohybrid composite

INTERVENTIONS:
Procedure: Zirconomer — zirconia modified glass ionomer
  Arms: Zirconomer in Class II cavities
Procedure: Nanohybrid composite — conventional composite
  Arms: Nanohybrid composite in Class II cavities

SUMMARY:
To achieve an optimal contact area is essential to avoid tooth migration, food impaction, and the occurrence of secondary caries. However, proximal restorations constitute challenge for the professional and tight contact points are difficult to obtain depending not only on tools used, but also on type of restorative material. Current tooth-colored restorative materials are not condensable and there is shrinkage with setting. The aim of this study is to compare the proximal contact tightness of zirconia reinforced glass ionomer versus conventional nanohybrid resin composite when used in class II cavities.

ELIGIBILITY:
Eligibility Criteria of participants:

Inclusion Criteria of participants:

* Patients with occlusoproximal caries in molars classified as ICDAS III or IV.
* 19-35 years.
* Males or Females.
* Co-operative patients approving to participate in the trial.

Exclusion criteria of participants:

* Pregnancy.
* Disabilities.
* Systemic disease or severe medical complications.
* Allergic history concerning methacrylate.
* Rampant caries.
* Heavy smoking.
* Xerostomia.
* Lack of compliance.
* Evidence of severe bruxism, clenching, or temporomandibular joint disorders.

  b- Eligibility Criteria of teeth:

Inclusion Criteria of teeth:

* Occlusoproximal caries in molars classified as ICDAS III or IV.
* Vital upper or lower posterior teeth with no signs of irreversible pulpitis.
* Intact contact with opposing teeth.
* Teeth with no previous restorations in other surfaces.

Exclusion criteria of the teeth:

* Extensive carious lesions
* Periapical pathology or signs of pulpal pathology.
* Tooth hypersensitivity.
* Possible prosthodontic restoration of teeth.
* Heavy occlusion and occlusal contacts or history of bruxism.
* Sever periodontal affection.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-09-12 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Contact Tightness | baseline, 3 months, 6 months, 9 months and 1 year
  Measuring the adequacy of proximal contact restoration using intervention ' zirconomer" versus control which is Nanohybrid resin composite.
  Heaviness of this contact using Modified USPHS criteria. USPHS criteria are standardized in which a dental floss is used.
  Contact tightness can have one of three scores:
  Alpha Bravo Charlie

CONTACTS AND LOCATIONS:
Overall Officials: Alaa F Abdelsalam, phD, Principal Investigator — lecturer of conservative dentistry, Cairo university; Hadier M Gad, PhD, Principal Investigator — Lecturer of conservative dentistry, Cairo university; Manar A Elmokanen, PhD, Principal Investigator — Lecturer of conservative dentistry, Cairo University
Locations (1):
- Faculty of dentistry Cairo university, Cairo, Manyal, Egypt

IPD SHARING:
Plan to Share IPD: No